CLINICAL TRIAL: NCT03601819
Title: Phase Ib, Open Label, Single Center Study of Pacritinib in Relapsed/Refractory Lymphoproliferative Disorders
Brief Title: Pacritinib in Relapsed/Refractory Lymphoproliferative Disorders
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2018.048; HUM00144759 (Other: University of Michigan)
Record Dates: First submitted 2018-07-18; First posted 2018-07-26 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell, Peripheral; Chronic Lymphocytic Leukemia; Lymphoproliferative Disorders; Waldenstrom Macroglobulinemia; Lymphoplasmacytic Lymphoma; Mantle Cell Lymphoma
Keywords: Relapsed; Refractory; MyD88; JAK2; JAK3; TYK2; IRAK1; CLL; SMZL; LPL; WM; MCL; CTCL; PTCL
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell, Peripheral; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoproliferative Disorders; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Recurrence | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pacritinib (Experimental): 200 mg twice daily (with possible dose reduction to 100 mg twice daily)
  Interventions: Drug: Pacritinib

INTERVENTIONS:
Drug: Pacritinib — Patients will receive continuous treatment until progressive disease, toxicity, or until any other condition for treatment discontinuation has been met.

SUMMARY:
This trial will determine the safety and tolerability of Pacritinib in patients with relapsed/refractory lymphoproliferative disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any of the following:

  1. Relapsed/refractory cutaneous (stage IIb-IV by ISCL/EORTC staging criteria) or peripheral T-cell lymphoma with progression after the last line of therapy and refractory to/intolerant of or have a contraindication to all established therapies known to provide clinical benefit (including brentuximab vedotin for patients with anaplastic large cell lymphomas) OR
  2. Chronic lymphocytic leukemia (CLL), splenic marginal zone lymphoma (SMZL), Waldenstrom's macroglobulinemia (WM)/lymphoplasmacytic lymphoma (LPL) or mantle cell lymphoma (MCL) with disease progression on ibrutinib or who discontinue ibrutinib due to toxicity/intolerance. In addition, patients should be refractory to/intolerant of or have a contraindication to all established therapies known to provide clinical benefit OR
  3. Any lymphoproliferative disorder who have failed at least 2 prior therapies and are refractory to/intolerant of or have a contraindication to all established therapies known to provide clinical benefit and have had mutational analysis or sequencing studies performed in a CLIA certified laboratory demonstrating a mutation or gene fusion involving MyD88, JAK2, JAK3, TYK2, or IRAK1 that are known or suspected to be "activating" (gain-of-function).
* Age ≥ 18 at time of enrollment
* ECOG ≤ 2 (Eastern Cooperative Oncology Group scoring system used to quantify general well-being and activities of daily life; scores range from 0 to 5 where 0 represents perfect health and 5 represents death.)
* Adequate organ and marrow function as defined in the protocol
* Ability to take oral medication without crushing, dissolving or chewing tablets.
* In the investigator's opinion, the patient requires immediate treatment.
* Ability to understand and the willingness to sign a written informed consent.
* In the investigator's opinion, the patient has the ability to communicate satisfactorily with the investigator and the study team, to participate fully in the study, and comply with all requirements.

Exclusion Criteria:

* History of, or a concurrent, clinically significant illness, medical condition or laboratory abnormality that, in the investigator's opinion, could affect the conduct of the study
* Pregnant or breast feeding women
* Unwilling or unable to use a medically acceptable form of contraception during the time of participation in the trial (sexual abstinence is permissible) unless documented successful vasectomy, hysterectomy, bilateral oophorectomy or post-menopausal for at least 2 years
* Uncontrolled current illness, including, but not limited to the following: Ongoing or active infections requiring intravenous antimicrobials; symptomatic congestive heart failure defined as NYHA class II, III or IV (Appendix II); unstable angina pectoris within 6 months of study enrollment; unstable cardiac arrhythmia; history of myocardial infarction, stroke or intracranial hemorrhage within 6 months prior to enrollment; moderate to severe hepatic impairment (Child-Pugh class B or C); psychiatric illness or social situations that would limit compliance with study requirements
* Known HIV infection
* Known positive Hepatitis B surface antigen or Hep C virus
* Recent (within 21 days of initiation of therapy, day 1) major surgery
* Less than 14 days have elapsed since last radiation therapy or chemotherapy treatment or patient has not recovered from all clinically significant treatment-related toxicity; less than 90 days have passed since date of autologous stem cell transplant and patient has not recovered to ≤grade 1 toxicity related to this procedure
* Use of systemic steroids (oral, inhaled, nasal, topical) at a dose less > 10 mg/day of prednisone
* Prior treatment with pacritinib
* Uncontrolled autoimmune hemolytic anemia (AIHA) or autoimmune thrombocytopenia (ITP). Coombs positivity in absence of hemolysis is not an exclusion.
* Requires anticoagulation with heparin, warfarin or equivalent Vit K antagonist
* History of significant bleeding (≥Grade 2 by CTCAE) history or complications (including bleeding that may have occurred while on ibrutinib)
* Hypersensitivity or allergic reaction to compounds related to pacritinib
* Treatment with potent CYP450 inducers and strong CYP3A4 inhibitors for which no alternative is available; treatment with strong CYP450 inducers or strong CYP3A4 inhibitors within 2 weeks of initiation of therapy, day 1
* Concurrent administration of QTc prolonging agents; significant QTc prolonging agents must be stopped within 5 half-lives of day 1.
* Any gastrointestinal or metabolic condition that could interfere with the absorption of oral medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-03-07 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities (DLT) | At 28 days
  Dose limiting toxicity (DLT) rate during the 1st cycle (28 days) of pacritinib.

SECONDARY OUTCOMES:
The proportion of patients that respond to treatment | Up to 2 years
  Overall response rate (ORR), defined as best disease response recorded from first day of treatment until disease progression or initiation of new antineoplastic therapy.
  Responses for patients with NHL or small lymphocytic lymphoma will be performed in accordance with the Revised Lugano classification staging system for non-Hodgkin's Lymphoma. Responses for patients with CLL will be evaluated in accordance with criteria of the International Workshop on Chronic Lymphocytic Leukemia, with the exception that lymphocytosis will not be the sole criteria for disease progression. Responses for CTCL will be assessed by the modified Severity Weighted Assessment Tool, response in blood, nodes, viscera, and the global composite scoring system.
The proportion of patients that experience a complete response (CR) | Up to 2 years
  Responses for patients with NHL or small lymphocytic lymphoma will be performed in accordance with the Revised Lugano classification staging system for non-Hodgkin's Lymphoma. Responses for patients with CLL will be evaluated in accordance with criteria of the International Workshop on Chronic Lymphocytic Leukemia, with the exception that lymphocytosis will not be the sole criteria for disease progression. Responses for CTCL will be assessed by the modified Severity Weighted Assessment Tool, response in blood, nodes, viscera, and the global composite scoring system.
Duration of response (DOR) | Up to 2 years
  DOR, defined as time from documented remission to the time of death, relapse, or initiation of alternative antineoplastic.
  Responses for patients with NHL or small lymphocytic lymphoma will be performed in accordance with the Revised Lugano classification staging system for non-Hodgkin's Lymphoma. Responses for patients with CLL will be evaluated in accordance with criteria of the International Workshop on Chronic Lymphocytic Leukemia, with the exception that lymphocytosis will not be the sole criteria for disease progression. Responses for CTCL will be assessed by the modified Severity Weighted Assessment Tool, response in blood, nodes, viscera, and the global composite scoring system.
Time to next treatment | Up to 2 years
  Time to next treatment, defined as time from first dose of pacritinib to initiation of alternative antineoplastic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Wilcox, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No